CLINICAL TRIAL: NCT03017937
Title: Sex and Age Ultrasound Response to Differential Jugular Vein Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-8580
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Concussion, Mild
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Q- collar (Experimental): All subjects will wear 3 sizes of the q-collar and ultrasound images of the jugular vein will be measured with each collar. Also, each subject will wear a pressure collar and ultrasound images of the jugular vein will be captured at each pressure point (0.1-0.5)
  Interventions: Device: Q-collar

INTERVENTIONS:
Device: Q-collar — capture ultrasound images at each pressure point

SUMMARY:
Clinical trials have suggested that this device is effective in mitigating changes in brain structure and function in athlete populations. The purpose of the current study is to measure the response of the jugular vein to various pressures applied by a generic compression device across various ages and gender. The relative jugular vein response will be measured using ultrasound.

DETAILED DESCRIPTION:
The Device has the promise of providing a novel mechanism for reducing or preventing the likelihood of TBI, and may be used in conjunction with other protective equipment. TBI is the leading cause of death in individuals under age 45. The cost of TBI in the U.S. is estimated at anywhere from $50 to $150 billion, annually. Concussion in female high school soccer players have been noted to occur at a rate of 4.5 concussions per 10,000 athletic exposures (Comstock, Currie et al. 2015). The investigators propose that Slosh Theory can explain these differences offering a mechanistic approach that could help shed light on further ways to alleviate the TBI burden on society. Note that Slosh Theory teaches that hydrodynamics (fluids moving within moving containers) contribute to, or are even the main etiology for, energy absorption of the cranial contents and that mitigation of SLOSH (increased compensatory reserve volume) may mitigate TBI. Significant morbidity, mortality, and related costs are caused by traumatic brain injury (TBI). A simple, effective, and lightweight device worn by athletes or war fighters in the field, designed to mitigate TBI resulting from blast trauma or concussive events, would save lives, and the huge costs currently being experienced for life-treatment of surviving victims. An externally-worn medical device (the Device) that applies mild jugular vein compression according to the principle of the Queckenstedt Maneuver, is being developed by Q30 Sports Science, LLC (Q30). Preliminary research suggests that the Device has the potential to reduce the likelihood of TBI. The currently developed collar (Smith 2009, Smith and Fisher 2011, Smith and Fisher 2011, Smith 2012) has been approved for studies in humans (IRB 2013-2240) and the results indicate safety for use during high demand and maximal exertion activities. Regarding safety, the externally worn collar is meticulously designed to mimic the body's own omohyoid muscle actions upon the jugular veins that will provide similar pressure and volume increases not to surpass that of a yawn or the mere act of just lying down. Initial safety testing and early clinical trials indicate that the collar application is both safe and efficacious to prevent brain microstructure and neurophysiological changes in response to head impacts.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy volunteer aged 7-60
* Able to provide written consent
* Able to tolerate hypercapnia for 1-2 minutes

Exclusion Criteria:

* Unable to provide written consent
* History of neurological deficits, previous cerebral infarction, or severe head trauma as indicated through pre-season screening:
* Medical contraindications to restriction of venous outflow via the internal jugular veins (known increased intracerebral pressure, metabolic acidosis or alkalosis)
* Glaucoma (Narrow Angle or Normal Tension)
* Hydrocephalus
* Recent penetrating brain trauma (within 6 months)
* Known carotid hypersensitivity
* Known increased intracranial pressure
* Central vein thrombosis
* Any known airway obstruction
* Any known seizure disorder

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 155 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Myer, PhD, Principal Investigator — Cincinnati Childrens Hospital
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Q- Collar
Started | 155
Completed | 155
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Q- Collar
Number analyzed (Participants) | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (14.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 86
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 155
Average neck size [Mean (Standard Deviation); unit: inches] | 13.5 (2.18)

OUTCOME MEASURES:

1. Primary Outcome: Neck Collar Size
Description: measurement of the neck collar size at each pressure level
Time Frame: 1 hour
Population: analysis broken down by gender and collar size
Measure: Mean (Standard Deviation); unit: inches
Groups:
- Females; Males: All subjects will wear 3 sizes of the q-collar and ultrasound images of the jugular vein will be measured with each collar. Also, each subject will wear a pressure collar and ultrasound images of the jugular vein will be captured at each pressure point (0.1-0.5)
  Q-collar: capture ultrasound images at each pressure point
Arm/Group | Females | Males
Number analyzed (Participants) | 69 | 86
inches
  Size 11 0.75: number analyzed (Participants) | 11 | 10
  Size 11 0.75 | 11.15 (0.052) | 11.11 (0.032)
  Size 11 1.0: number analyzed (Participants) | 11 | 10
  Size 11 1.0 | 11.25 (0.052) | 11.21 (0.032)
  Size 11 1.25: number analyzed (Participants) | 11 | 10
  Size 11 1.25 | 11.145 (0.052) | 11.11 (0.032)
  Size 12 0.75: number analyzed (Participants) | 16 | 9
  Size 12 0.75 | 12.25 (0.052) | 12.28 (0.044)
  Size 12 1.0: number analyzed (Participants) | 16 | 9
  Size 12 1.0 | 12.25 (0.052) | 12.22 (0.044)
  Size 12 1.25: number analyzed (Participants) | 16 | 9
  Size 12 1.25 | 12.25 (0.052) | 12.22 (0.044)
  Size 13 0.75: number analyzed (Participants) | 15 | 9
  Size 13 0.75 | 13.18 (0.10) | 13.23 (0.1)
  Size 13 1.0: number analyzed (Participants) | 15 | 9
  Size 13 1.0 | 13.18 (0.101) | 13.23 (0.1)
  Size 13 1.25: number analyzed (Participants) | 15 | 9
  Size 13 1.25 | 13.24 (0.051) | 13.27 (0.05)
  Size 14 0.75: number analyzed (Participants) | 9 | 9
  Size 14 0.75 | 14.133 (0.05) | 14.156 (0.053)
  Size 14 1.0: number analyzed (Participants) | 9 | 9
  Size 14 1.0 | 14.133 (0.05) | 14.167 (0.05)
  Size 14 1.25: number analyzed (Participants) | 9 | 9
  Size 14 1.25 | 14.167 (0.05) | 14.133 (0.05)
  Size 15 0.75: number analyzed (Participants) | 8 | 14
  Size 15 0.75 | 15.15 (0.053) | 15.14 (0.051)
  Size 15 1.0: number analyzed (Participants) | 8 | 14
  Size 15 1.0 | 15.2 (0.107) | 15.19 (0.103)
  Size 15 1.25: number analyzed (Participants) | 8 | 14
  Size 15 1.25 | 15.15 (0.053) | 15.14 (0.051)
  Size 16 0.75: number analyzed (Participants) | 8 | 13
  Size 16 0.75 | 16.26 (0.052) | 16.27 (0.05)
  Size 16 1.0: number analyzed (Participants) | 8 | 13
  Size 16 1.0 | 16.24 (0.052) | 16.23 (0.05)
  Size 16 1.25: number analyzed (Participants) | 8 | 13
  Size 16 1.25 | 16.23 (0.104) | 16.24 (0.1)
  Size 17 0.75: number analyzed (Participants) | 2 | 11
  Size 17 0.75 | 17.1 (0) | 17.15 (0.052)
  Size 17 1.0: number analyzed (Participants) | 2 | 11
  Size 17 1.0 | 17.2 (0) | 17.15 (0.052)
  Size 17 1.25: number analyzed (Participants) | 2 | 11
  Size 17 1.25 | 17.3 (0) | 17.19 (0.10)
  Size 18 0.75: number analyzed (Participants) | 0 | 11
  Size 18 0.75 |  | 18.15 (0.93)
  Size 18 1.0: number analyzed (Participants) | 0 | 11
  Size 18 1.0 |  | 18.15 (0.093)
  Size 18 1.25: number analyzed (Participants) | 0 | 11
  Size 18 1.25 |  | 18.13 (0.047)

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | Q- Collar
All-Cause Mortality (participants affected / at risk) | 0/155
Serious Adverse Events (participants affected / at risk) | 0/155
Other Adverse Events (participants affected / at risk) | 0/155

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT03017937/Prot_SAP_000.pdf
  • Informed Consent Form (2016-11-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT03017937/ICF_001.pdf